CLINICAL TRIAL: NCT05434572
Title: Center for Inherited Muscle Research Neuromuscular Research Biobank
Brief Title: CIMR Neuromuscular Research Biobank
Acronym: NRB-0001
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20021172
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Diseases; Neuromuscular Disorder; Neuromuscular Diseases in Children
Keywords: Neuromuscular; Research Repository; Biobank; Neuromuscular Disorder
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — As part of this repository, subjects will also have the option to allow a cell line to be made from their blood, muscle, or skin biopsies to provide a renewable supply of DNA and other cell components for research. A cell line is a frozen sample of specially processed cells from blood that allows us to grow more cells and obtain more DNA and other cell components, such as RNA or proteins, for future research. The cell line would not be labeled with the subjects name, address, birthdate, or other personal identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research repository is to collect, store, and share with other researchers any tissues that subjects with all types of neuromuscular disease are willing to donate. These samples will be stored at Virginia Commonwealth University (VCU) and will be used for future research with this population.

DETAILED DESCRIPTION:
The study involves collection of medical information about research participants and their families. No identifying information about family members will be collected. Research participants will be asked for any general knowledge they have related to possible neurological disorders.

Research participants are also given the opportunity to provide blood, skin cells, urine, saliva, fecal matter, muscle tissue, cells, DNA and/or RNA samples.

Before any study procedures take place, the informed consent form will be provided and reviewed with potential research participants in detail. Potential research participants will have an opportunity to ask additional questions before starting any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Positive diagnosis or suspected diagnosis of neuromuscular disease, or
* Family history of neuromuscular disease, or
* Healthy volunteer
* Age Neonates-75

Exclusion Criteria:

* Unwilling to sign consent

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a very inclusive study that will allow samples from known subjects of sites' neuromuscular clinics, associated family members, and healthy volunteers. This study will include subjects with any form of neuromuscular disorder, including neuromuscular disorders of unknown etiology.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
To collect, store, and share with other researchers any tissues that subjects with all types of neuromuscular disease are willing to donate. | Baseline
  Subjects will have the opportunity to provide the following samples: saliva or cheek swab, urine sample (up to 15ml), feces (up to 2mg of a stool sample), blood (up to 40ml), muscle biopsy tissue, and cell line (subjects have the option to allow a cell line to be made from their blood, muscle, or skin biopsies to provide a renewable supply of DNA and other cell components for research)

SECONDARY OUTCOMES:
To collect medical history information from subjects with all types of neuromuscular disease and healthy controls. | Baseline
  Information will be collected from the subject medical records and will include care they have received in the past, are receiving now, or may receive in the future. Subject information may include name, age, gender, diagnosis, and other medical history information that may be beneficial to the research staff.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided